CLINICAL TRIAL: NCT02785523
Title: Clinical Trial on Ganoderma Spore Lipids Combined With Chemo in Patients With G.I. Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaonan Cui (Other)
Responsible Party: Sponsor-Investigator, Xiaonan Cui, Professor, Chief Physician, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G20090400
Record Dates: First submitted 2016-03-25; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- G. SPORE LIPIDS (Experimental): Form: Capsule Dosage and frequency: This group receives ganoderma spore lipids capsules 600mg TID in addition to the chemotherapy.
  Duration: 6 chemotherapy cycles.
  Interventions: Drug: Ganoderma Spore Lipids; Drug: Chemotherapy
- Placebo (Placebo Comparator): Form: Capsule Dosage and frequency: This group receives placebo capsules 600mg TID in addition to the chemotherapy.
  Duration: 6 chemotherapy cycles.
  Interventions: Drug: Placebo; Drug: Chemotherapy

INTERVENTIONS:
Drug: Ganoderma Spore Lipids
  Other Names: G. SPORE LIPIDS
  Arms: G. SPORE LIPIDS
Drug: Placebo
  Arms: Placebo
Drug: Chemotherapy

SUMMARY:
A phase III double-blind randomized clinical trial on the effects of ganoderma spore lipids to the immunological response in patients with G.I. Cancers. The trial is randomized, double-blind. Cancer patients are diagnosed based on pathology or cell biology. Patients are randomized into 2 groups: both groups receive chemotherapy. Either group receives ganoderma spore lipids or placebo capsules 600mg three times a day (TID) in addition to the chemotherapy. Clinical evaluation includes chemotherapy drug toxicities, life quality improvement. Blood biochemistry tests mainly include malondialdehyde (MDA), superoxide dismutase (SOD), glutathione peroxidase (GSH-Px), adrenaline, nor-adrenaline, tumor necrosis factor (TNF)-α, interleukin (IL)-1b, interleukin (IL)-6, cell flow cytometry on Th1, Th2, Th17, Treg cytokines, as well as serum cortisol, estradiol (female), progesterone (female), testosterone (male), etc.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80, male and female.
* Diagnosis: imaging, cell and pathology report.
* Eastern Cooperative Oncology Group (ECOG) O-2, life expectancy more than 3 months.
* Chemotherapy is not contraindicated.
* No apparent surgical trauma during the previous 2 weeks.
* Past treatment:

  * Biological treatment: at least 4 weeks after previous treatment with immunotherapy or other biological; chemotherapy, at least 6 months after last treatment with chemotherapy and or target therapy.
  * Surgery: had not received transplantation surgery, at least 2 weeks after last major surgery.

Exclusion Criteria:

* A purulent and chronic infection of wound healing delayed.
* Diseases of the blood system.
* Abnormal blood coagulation function.
* Severe brain disease or primary brain tumors without control, and mentally ill person.
* Patients with brain metastases.
* Pregnant or lactating women.
* Patients (male/female) with fertility, But the patients themselves or their spouses do not take effective contraception.
* Allergic constitution.
* In addition, patients taking part in other clinical trials, being treated with other biotherapy or immunotherapy and researchers consider not suitable for clinical subjects for other reasons will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events: neutropenia, leukopenia, thrombocytopenia, anemia, nausea, vomit, fatigue, loss of appetite. | Cycle 2, cycle 4, cycle 6(each cycle is 21 days).
Assessing the quality of life(QOL) in 5 grades and recording: appetite, mental state, sleep, fatigue, pain, attitude towards treatment, daily life ability, treatment of severity of side effects. | Cycle 2, cycle 4, cycle 6(each cycle is 21 days).

SECONDARY OUTCOMES:
Th1/Th2, Th17/Treg in blood. | Cycle 2, cycle 4, cycle 6(each cycle is 21 days).
Interleukin(IL)-1b, interleukin(IL)-6, tumor necrosis factor(TNF)-α in blood. | Cycle 2, cycle 4, cycle 6(each cycle is 21 days).
Estradiol (female), progesterone (female), testosterone (male) in blood. | Cycle 2, cycle 4, cycle 6(each cycle is 21 days).
Vanillylmandelic acid (VMA) in urine. | Cycle 2, cycle 4, cycle 6(each cycle is 21 days).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD, PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided